CLINICAL TRIAL: NCT03618147
Title: Kuwait National Primary Immunodeficiency Registry (KNPIDR)
Brief Title: Primary Immunodeficiency in Kuwait
Status: Completed | Type: Observational
Sponsor: Kuwait Society for Allergy and Clinical Immunology (Other)
Responsible Party: Principal Investigator, Waleed Al-Herz, Associate Professor of Pediatrics, Kuwait Society for Allergy and Clinical Immunology
Other Study IDs: IIR - K W T - 0 0 2 0 7 1
Record Dates: First submitted 2018-07-30; First posted 2018-08-07 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Background/Rationale: Epidemiological data about Primary Immunodeficiency Disorders (PIDD) in Kuwait is needed to better understand peculiarities and to compare them with other regions and ethnicity.
* Study hypothesis: PIDD is relatively common in Kuwait compared to populations from different geographic areas. The distribution of PIDD in Kuwait is different from other geographic areas with more severe forms being more frequent.
* Brief inclusion and exclusion criteria of study participants: PIDD patients presented at different clinics/hospital in Kuwait. Patients with secondary immunodeficiencies (drug induced, virus induced, and immunodeficiency associated with metabolic disorders... ect), will be excluded
* Estimated sample size of the study: All patients who were registered in KNPIDR since 2004 will be included in the study along with the new patients who will be recruited during the study period.
* Primary objectives:

  * Determine the prevalence and frequency of different PIDD in Kuwait
  * Identify clinical presentation patterns for PIDD in Kuwait
  * Identify natural history of PIDD in Kuwait
  * Help to asses epidemiology of PIDD in Kuwait
  * Determine particularities about PIDD affecting the population in Kuwait
  * Determine the health impact of PIDD in Kuwait
  * Development of strategies to improve the care and the quality of life of patients with PIDD

ELIGIBILITY:
Inclusion Criteria:

* PIDD patients presented at different clinics/hospital in Kuwait
* Exclusion Criteria: Patients with secondary immunodeficiencies (drug induced, virus induced, and immunodeficiency associated with metabolic disorders... ect)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PIDD patients in Kuwait
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Deprtmemt, Alsabah hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PID Patients: All patients who were diagnosed with primary immunodeficiency
Period: Overall Study
Arm/Group | PID Patients
Started | 314
Completed | 314
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All PID patients
Groups:
- PID Arab Patients: All patients diagnosed with PID
Arm/Group | PID Arab Patients
Number analyzed (Participants) | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 295
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149
  Male | 165
Race/Ethnicity, Customized [Number; unit: participants] — All patients are Arab
  participants
    Arab patients | 314

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Different Epidemiological Features
Time Frame: 15 years
Population: PID patients
Measure: Number; unit: patients
Arm/Group | PID Patients
Number analyzed (Participants) | 314
patients
  Kuwaiti patients | 287
  immunodeficiencies affecting cellular and humoral | 100
  combined immunodeficiencies with associated syndro | 68
  predominantly antibody deficiencies | 56
  diseases of immune dysregulation | 47
  Phagocytic defects | 20
  autoinflammatory disorders | 1
  Complement deficiencies | 22
  Parental consanguinity | 245
  Family history of PID | 157
  Genetic testing | 217
  IVIG treatment | 175
  Stem cell transplant | 72
  Deaths | 81

2. Primary Outcome: Number of Overall and New Cases of PID Per 100,000 Kuwaitis
Time Frame: 15 years
Measure: Number; unit: Cases per 100,000 Kuwaiti
Groups:
- PID Patients: PID Arab patients
Arm/Group | PID Patients
Number analyzed (Participants) | 314
Cases per 100,000 Kuwaiti
  Overall Cases | 20
  New Cases | 25

ADVERSE EVENTS:
Time Frame: 15 years
Description: Serious Adverse Events and Other (Not Including Serious) Adverse Events" were not monitored/assessed
Arm/Group | PID Patients
All-Cause Mortality (participants affected / at risk) | 81/314
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PID Patients (N=0)
(General disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03618147/Prot_000.pdf